CLINICAL TRIAL: NCT05417334
Title: Effect of Radiofrequency in the Treatment of de Novo Dyspareunia at 4 to 16 Months Postpartum: Randomised Prospective Trial
Brief Title: Effect of Radiofrequency in the Treatment of de Novo Dyspareunia at 4 to 16 Months Postpartum.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carla Box, Physical Therapist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCB/2020/0484
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dyspareunia
Keywords: dyspareunia; radiofrequency; postpartum pain; perineal massage; episiotomy
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ON Radiofrequency treatment (Active Comparator): Application of the technique in the intervention group (activated resistive capacitive monopolar radiofrequency therapy): the intervention group will receive treatment with activated RF, with the electrode at a medium intensity for 20 minutes per session during a total of 5 sessions, the 3 first ones held weekly and the 2 last ones every other week.
  Interventions: Device: Resistive Capicitive Monopolar Radiofrequency
- Sham Radiofrequency treatment (Sham Comparator): Application of the technique in the intervention group (inactive resistive capacitive monopolar radiofrequency therapy): the intervention group will receive treatment with inactive RF, with the electrode at a medium intensity for 20 minutes per session during a total of 5 sessions, the 3 first ones held weekly and the 2 last ones every other week.
  Interventions: Device: Resistive Capicitive Monopolar Radiofrequency

INTERVENTIONS:
Device: Resistive Capicitive Monopolar Radiofrequency — 5 Radiofrequency sessions including the abdominal region, the vulva and pelvic floor tissue and Thiele massage done daily by the patient at home

SUMMARY:
This study evaluates if the application of resistive capacitive monopolar radiofrequency therapy associated with Thiele massage is effective when treating de novo dyspareunia at 4 to 9 months postpartum.

DETAILED DESCRIPTION:
Dyspareunia is a type of genito-pelvic pain (GPP) that takes place during vaginal penetration at some point in sexual intercourse. It greatly affects quality of life as well as psychological and sexual wellbeing. A delivery with episiotomy, perineal tearing or labor dystocia using forceps or vacuum, are risk factors that contribute to the appearance of de novo dyspareunia with a prevalence of 17-45% at 6 months postpartum.

There is no evidence in the scientific literature of the effect of radiofrequency is this group of patients, however there is a clinical trial that describes the effect in scar tissue although not in the perineum. It is for all of the above that the following project is proposed, to evaluate the effect of RF in perineal healing and vaginal trigger points caused as a consequence of GPP.

The main objective of this study is to evaluate the role that radiofrequency (RF) plays in reducing the level of pain in de novo dyspareunia in postpartum women that persists from 4 to 9 months.

ELIGIBILITY:
Inclusion Criteria:

* 4-9 postpartum
* de novo dyspareunia after delivery
* obstetric injury
* Grant informed consent

Exclusion Criteria:

* radiofrequency contraindications (pacemaker, active infection or pregnancy)
* cesarean section
* dyspareunia previous to labour
* previous vulvo-vaginal pathology
* patients with postpartum depression
* patients with a pelvic region oncological history

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postpartum women
Enrollment: 110 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change of the baseline Level of pain during penetration and after 5 sessions | Baseline and after 7 weeks
  Using the Visual Analogue Scale (VAS), where 10 is the highest level of pain possible and 0 is no pain at all.

SECONDARY OUTCOMES:
Change of the baseline Sexual function and after 5 sessions | Baseline and after 7 weeks
  Using the Female Sexual Function Index (FSFI), where higher scores indicate higher degrees of sexual functioning of a total of 36 points (and lower pain).
Change of the baseline muscle pain points and after 5 sessions | Baseline and after 7 weeks
  A physical evaluation held by the physical therapist seeking for pain points and asking the patient to score the amount of pain using the visual analogue scale (VAS) where 10 is the highest level of pain possible and 0 is no pain at all.
Change in Pelvic floor dysfunctions in the baseline assesment and after 5 sessions | Baseline and after 7 weeks
  Using the Pelvic Floor Distress Inventory-20 questionnaire (PFDI-20), in which the higher the score the greater the perceived impact that the pelvic floor dysfunction has on the patient's life (range 0 to 300 points).
Change of the baseline affection on the quality of life and after 5 sessions | Baseline and after 7 weeks
  Using the EuroQuality of life-5D (EQ5D),where the maximum score of 1 indicates the best health state and therefore, higher scores indicate more severe or frequent problems (range from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No